CLINICAL TRIAL: NCT06158503
Title: GLYcemic COntrol and OSTEOhealth: Impact of Short-Term Glycemic Control on Skeletal Outcomes in Adults With Type 1 Diabetes
Brief Title: Glycemic Control and Osteohealth in Adults Living With Type 1 Diabetes
Acronym: GLYCO-OSTEO
Status: Recruiting | Type: Observational
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Laval University (Other); Institut de Recherches Cliniques de Montreal (Other)
Responsible Party: Principal Investigator, Rémi Rabasa-Lhoret, Co-investigator, Centre hospitalier de l'Université de Montréal (CHUM)
Other Study IDs: MP-02-2024-11708
Record Dates: First submitted 2023-11-28; First posted 2023-12-06 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 Diabetes; Bone Health; Automated Insulin Delivery
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insemination, Artificial, Heterologous

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples before and after initiation of the AID system.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- AID initiation: The participants will be selected on the basis that they are planning to start using one of the commercially available AID.
  They will start treatment after the initial measurements (baseline), then repeat the measurements at 2 and 4 months post-AID.
  Interventions: Device: AID

INTERVENTIONS:
Device: AID — Initiation of an automated insulin delivery system

SUMMARY:
Bone damage is frequently observed in type 1 diabetes, and hyperglycemia is associated with an increased risk of fracture. This pilot study in 25 people living with type 1 diabetes aims to determine whether the introduction of an automated insulin delivery (AID) system improves bone markers through rapide optimization of glycemic control. Measurements will be taken before the start of AID, 2 months and 4 months afterwards.

DETAILED DESCRIPTION:
Background: Bone damage is a frequently overlooked complication of type 1 diabetes (T1D), but significantly increases the risk of fractures as early as childhood. Fractures in individuals with T1D increase the risk of delayed healing, postoperative complications, loss of autonomy, reduced quality of life and even mortality. The pathophysiology of bone alterations in T1D probably differs from that of primary osteoporosis. Studies show lower bone mineral density in T1D, but this is not sufficient to fully explain the risk of fractures. T1D is also characterized by low bone remodeling and altered bone microarchitecture. Although chronic hyperglycemia is a risk factor for fracture in T1DM, the effect of improved glycemic control on bone markers remains unclear. The main hypothesis is that rapid optimization of the glycemic profile (hyperglycemia and variability) may improve bone remodeling in people living with T1DM who have suboptimal glycemic control.

Aim: The primary objective of this pilot study is to quantify the proportion of participants significantly increasing at least one of the serum markers of bone remodeling post-installation of an automated insulin delivery system.

Secondary objectives are to quantify: 1) the magnitude of change in each of the serum markers of bone remodeling pre-intervention and at 2 and 4 months post-intervention; 2) the efficacy of the automated insulin delivery system in terms of glycemic control and variability (mean change in HbA1c and glycemic parameters derived from the continuous glucose monitoring system).

Methods: method: This is a prospective pilot study involving 25 adults aged 18 and over living with T1DM or latent autoimmune diabetes of adults (LADA) who are interested in starting an automated insulin delivery system (artificial pancreas).

This study will involve 3 visits:

1. Visit 1: before installation of the automated insulin delivery system,
2. Visit 2: follow-up at 2 months after installation of the automated insulin delivery system,
3. Visit 3: follow-up at 4 months after installation of the automated insulin delivery system.

During visits 1 and 3, participants will take a blood sample, perform a brief physical examination and complete questionnaires.

During visit 1, participants will also undertake a urine sample, and the research team will conduct a brief interview to obtain information on their diabetes diagnosis, associated complications, and medication use.

During Visit 2: blood sample only.

The project will not interfere with the participant's diabetes management. They will be asked to share a copy of their 14-day continuous glucose monitoring profile during the visit periods.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Diagnosis of T1D or latent autoimmune diabetes of adults (LADA) for at least one year;
* Current HbA1c >8.0% and high glycemic variability (CV >36.0% using CGM);
* Participant planning to start using one of the commercially available AID;
* Anticipated use of the closed-loop mode;
* Willing to share CGM data during the study period.

Exclusion Criteria:

* Woman who was pregnant, gave birth or breastfed less than 6 months before the beginning of the study or who plans to become pregnant during the study;
* Conditions affecting bone turnover markers, such as chronic kidney disease (estimated GFR <30 ml/min), liver disease, intestinal malabsorption including celiac disease, organ transplant, active cancer, rheumatoid arthritis, and endocrinopathies (active hyperthyroidism, uncontrolled hypothyroidism with abnormal TSH, parathyroid disease, hypogonadism, Cushing syndrome, adrenal insufficiency and acromegaly);
* Anticipated therapeutic change and/or type of CGM sensor, insulin pump, or AID during the study period;
* Anticipated need to use acetaminophen during the study period at a dose above 1g every 6 hours;
* Current or anticipated use of hydroxyurea;
* Intake in the past 12 months of drugs influencing bone turnover markers, such as oral or intra-articular glucocorticoids (≥ 7.5 mg daily Prednisone or equivalent during ≥ 3 months or ≥ four intra-articular glucocorticoid infiltrations in the past year), aromatase inhibitor therapy for breast cancer and anti-androgen therapy for prostate cancer, anticoagulants, SGLT-2 inhibitors, thiazolidinediones, and anti-osteoporosis drugs;
* Unable to consent.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People living with type 1 diabetes who do not use an automated insulin delivery system but wish to do so. The study takes place around the initiation of AID.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Bone remodeling improvement | 4 months
  The proportion of participants increasing at least one of the serum bone turnover markers above the least significant change (>43% for CTX, >25.49% for procollagen type 1 N-terminal propeptide (P1NP) and >25.65% for osteocalin).

SECONDARY OUTCOMES:
Carboxy-terminal collagen crosslinks change | 2 months
  Magnitude of the change and the variance for CTX
Carboxy-terminal collagen crosslinks change | 4 months
  Magnitude of the change and the variance for CTX
N-terminal propeptide (P1NP) change | 2 months
  Magnitude of the change and the variance for P1NP
N-terminal propeptide (P1NP) change | 4 months
  Magnitude of the change and the variance for P1NP
Osteocalin change | 2 months
  Magnitude of the change and the variance for Osteocalin
Osteocalin change | 4 months
  Magnitude of the change and the variance for Osteocalin
HbA1c change | 2 months
  Mean change of glycated hemoglobin (HbA1c)
HbA1c change | 4 months
  Mean change of glycated hemoglobin (HbA1c)

CONTACTS AND LOCATIONS:
Overall Officials: Rémi Rabasa-Lhoret, MD, PhD, Principal Investigator — IRCM
Locations (2):
- Canada (2):
  - CHUM, Montreal, Quebec
  - Centre Hospitalier de l'Université de Montréal, Montreal